CLINICAL TRIAL: NCT05663983
Title: Valutazione Retrospettiva Multicentrica e Risultati Delle Strategie Terapeutiche Nei Pazienti Adolescenti o Giovani Adulti (AYA). Studio di Collaborazione Fra AIEOP e FIL
Brief Title: Multicentric and Retrospective Analysis of Adolescent Young Adult (AYA) Hodgkins' Lymphoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Campus Bio-Medico University (Other)
Collaborators: Associazione Italiana di Ematologia e Oncologia Pediatrica (Unknown); Fondazione Italiana Linfomi (Unknown)
Responsible Party: Principal Investigator, Luigi Rigacci, Clinical Trial Office Campus Bio-Medico, Campus Bio-Medico University
Other Study IDs: AYA
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Hodgkin Lymphoma; Adolescent Behavior; Chemotherapy Effect
MeSH Terms: conditions — Hodgkin Disease; Adolescent Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIEOP: This is a National Association for the treatment of pediatric patients with hematological or oncological disease
  Interventions: Behavioral: Description of therapeutical results
- FIL: This is a National Association that brings together many centers with particular attention to the treatment of adult lymphomas
  Interventions: Behavioral: Description of therapeutical results

INTERVENTIONS:
Behavioral: Description of therapeutical results — Comparison between two groups of patients treated in different realities (Pediatric Hospital or Adult General Hospital)

SUMMARY:
The principal aim of this study is to collect retrospectively all Adolescent Young Adult patients affected by Hodgkin's Lymphoma and treated in pediatric or adult haemato-oncology Centers. The data set collection aims to define the therapy performed and the results obtained in terms of overall survival and acute or late complications.

DETAILED DESCRIPTION:
Hodgkin lymphoma (HL) represents approximately 0.5% of cancer diagnosis each year in developed countries (1, 2). This translates to an annual incidence of 8500 individuals per year in the United States and an incidence rate of 2.49 per 100.000 lymphoid malignancies in Europe (2, 3). A classical bimodal distribution is reported with a first peak occurring in patients between the ages of 15 and 30 years and a second peak in those older than 55 years (4). HL is one of the most common malignancies to occur in the adolescent and young adult (AYA) population. This population is defined by the National Cancer Institute as people diagnosed with cancer between the ages of 15 and 39 years.

The choice of therapy for AYA patients is typically determined by the treatment setting and referral patterns. Patients who are younger than 18 years are usually referred to pediatric Centers, where many patients are treated in the context of clinical trials. For patients treated by adult haematologists many are treated in the community setting.

Considerable variability exists between the treatment of adult and pediatric patients, including the choice of chemotherapeutic agents and the role of radiation. In both the pediatric and adult settings there has been increasing focus on balancing the risk of relapse with the risk of secondary side effects. De-intensification for low-risk patients using PET-adapted strategies is a modern approach that has been applied to all patients with HL independent of age. Variability among age groups still results in uncertainty regarding the optimal treatment approach in the AYA population.

This is a retrospective observational study involving Italian Centers that treat adolescents and young adults Hodgkin lymphoma patients. This type of patients can be treated either in a Pediatric Institution or in Adult Institution with different supportive and therapeutical approaches.

The primary objectives will be overall survival according to different treatment. Secondary end points will be acute or late complications comparing different treatments choice in an homogeneous group of patients, progression free survival according to different treatment.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with diagnosis of Hodgkin Lymphoma with an age at diagnosis ranging between 15 and 24 years enrolled in prospective studies either in AIEOP group and in FIL group or patients treated consecutively in single centers affiliated to AIEOP or FIL and registered in single institutional data base.
* All Hodgkin subtype

Exclusion Criteria:

* None

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a retrospective observational study involving Italian Centers that treat adolescents and young adults Hodgkin lymphoma patients. This type of patients can be treated either in a Pediatric Institution or in Adult Institution with different supportive and therapeutical approaches.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival according to different treatment. | 2004 to 2016
  To evaluate if there are differences in treatment of pediatric or adult subset of patients

SECONDARY OUTCOMES:
Acute or late complications | 2004 to 2016
  Comparing different treatments choice in an homogeneous group of patients
Progression free survival | 2004 to 2016
  According to different treatment

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR